CLINICAL TRIAL: NCT02650323
Title: Registro Campano Delle Sindromi Coronariche Acute
Brief Title: Observational Registry on Acute Coronary Syndromes in Campania
Acronym: Campania RESCA
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruno Trimarco, Director of Cardiology, Federico II University
Other Study IDs: 216_2105
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This registry aims to collect data related to management of patients affected by acute coronary syndromes and hospitalized in the Campania Region of Italy

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for acute coronary syndromes

Exclusion Criteria:

* Refuse to provide informed consent for study enrollment

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patints hospitalized for Acute Coronary Syndromes
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, MD, Study Chair — University of Napoli Federico II; RAFFAELE IZZO, Study Director — Federico II University
Locations (1):
- Ambulatorio Ipertensione e Unità Coronarica Federico II University, Napoli, Italy